CLINICAL TRIAL: NCT03141918
Title: Effect of Supplementation of Bioactive Compounds on the Energy Metabolism of People Living With HIV / AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, TATIANE ANDREZA LIMA DA SILVA, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: COMPOSTOS_BIOATIVOS_VIVER MAIS
Record Dates: First submitted 2017-02-23; First posted 2017-05-05 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Curcumin group 1 (Experimental): Intervention will be with intake of curcumin, 1000mg per 30 days
  Interventions: Dietary Supplement: Curcumin
- Curcumin group 2 (Placebo Comparator): Intervention will be with placebo intake of curcumin, 1000mg per 30 days
  Interventions: Other: Placebo of Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin — The intervention will consist of the supplementation of curcumin for 30 days. Curcumin supplementation will be done by administration of 2 doses of 500mg of the product BioMor Curcumin® which is composed of 95% standardized extract of the root extract of Curcuma longa.
  Arms: Curcumin group 1
Other: Placebo of Curcumin — The intervention will consist of the placebo administration curcumin for 30 days.
  The Curcumin placebo will be given in 2 doses of 500mg per day.
  Arms: Curcumin group 2

SUMMARY:
Among the many changes associated with the impact of HIV and the long-term use of antiretroviral therapy, metabolics are important because they are important risk factors for the development of cardiovascular diseases. The objective of the present study is to evaluate the effect of the supplementation of curcumin, on the oxidation of resting energetic substrates in HIV / AIDS patients. The sample will be composed of adults living with HIV / AIDS on antiretroviral therapy for at least 6 months. Supplements will be made separately for 30 days and will be evaluated before and after the intervention the following parameters: body composition, energy metabolism, biochemical parameters and a structured anamnesis. Food consumption and the level of physical activity of the volunteers will be controlled.

DETAILED DESCRIPTION:
The study is characterized as a double-blind randomized clinical trial. Participants in the study will be adults living with HIV / AIDS who undergo regular clinical follow-up at some Specialized HIV / AIDS Care Service.

The sample will consist of 20 volunteers, 10 in the experimental group (GE) and 10 in the control group (CG). Participants will be randomly assigned to one of the groups by lottery by a researcher not participating in the study. The researcher responsible, as well as the volunteers, will not be aware of which participants are in the GE or the GC.

The study will be carried out in the Movement Laboratory of the Physical Education Department of the Federal University of Rio Grande do Norte.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral therapy has been available for at least 6 months, aged 18 years or over.

Exclusion Criteria:

* Individuals with endocrine and pregnant disorders will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
The oxidation of energetic substrates evaluation at rest | 10 DAYS
  The oxidation of energetic substrates evaluation at rest will be performed by indirect calorimetry, a gold standard method for the measurement of energy expenditure, making feasible through the breath by breath technique, weightings to quantify the Caloric expenditure from oxidation fats and carbohydrates. Evaluation will not offer any discomfort since the volunteer will lie flat without moving with a mask fixed on his face, which picks up the breathed and expired gases to be measured by the Respiratory Analyzer - Metalyzer 3B-MICROMED®.
  To determine oxidation of energetic substrates, subjects will be instructed to sleep approximately for 8 hours the night before, to fast for 12 hours, not to exercise and not to drink caffeinated beverages or alcohol in the 24 hours before the test. Such care should be taken in order to reduce the influence of the thermal effect of food and physical activity on resting metabolism

SECONDARY OUTCOMES:
Energy expenditure at rest | 10 DAYS
  The evaluation of resting energy expenditure will be performed by indirect calorimetry, a gold standard method for the measurement of energy expenditure, making feasible through the breath by breath technique, weightings to quantify the energy expenditure of rest. Evaluation will not offer any discomfort since the volunteer will lie flat without moving with a mask fixed on his face, which picks up the breathed and expired gases to be measured by the Respiratory Analyzer - Metalyzer 3B-MICROMED®.
  To determine resting energy expenditure, subjects will be instructed to sleep approximately for 8 hours the night before, to fast for 12 hours, not to exercise and not to drink caffeinated beverages or alcohol in the 24 hours before the test. Such care should be taken in order to reduce the influence of the thermal effect of food and physical activity on resting metabolism.
The glycemia evaluation | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature. Serum levels of glucose will be performed by enzyme-colorimetric assays using Labtest Diagnostic kits suitable for the RA-50 semi-automated biochemical analyzer (Bayer Diagnostics Chemistry System, Dublin).
The insulin evaluation | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature.Serum levels of insulin will be performed by enzyme-colorimetric assays using Labtest Diagnostic kits suitable for the RA-50 semi-automated biochemical analyzer (Bayer Diagnostics Chemistry System, Dublin).
The total cholesterol evalution | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature.Serum levels of total cholesterol will be performed by enzyme-colorimetric assays using Labtest Diagnostic kits suitable for the RA-50 semi-automated biochemical analyzer (Bayer Diagnostics Chemistry System, Dublin).
The LDL cholesterol evalution | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature.Serum levels of LDL cholesterol will be performed by enzyme-colorimetric assays using Labtest Diagnostic kits suitable for the RA-50 semi-automated biochemical analyzer (Bayer Diagnostics Chemistry System, Dublin).
The HDL cholesterol evalution | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature.Serum levels of HDL cholesterol will be performed by enzyme-colorimetric assays using Labtest Diagnostic kits suitable for the RA-50 semi-automated biochemical analyzer (Bayer Diagnostics Chemistry System, Dublin).
The triglycerides evalution | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature.Serum levels of triglycerides will be performed by enzyme-colorimetric assays using Labtest Diagnostic kits suitable for the RA-50 semi-automated biochemical analyzer (Bayer Diagnostics Chemistry System, Dublin).
The inflammatory markers evalution | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature.
The oxidative stress markers evalution | 10 DAYS
  Individuals will undergo a peripheral vein puncture in the morning after fasting from 12 to 14 h. Blood will be collected in 30 ml of blood in vacuum containment tubes without anticoagulant; Tubes will be identified with a different registration number for each participant.In order to obtain the serum, the blood samples will be centrifuged for 10 min at 2500 rpm at room temperature.

OTHER OUTCOMES:
Body composition | 10 DAYS
  The body composition will be evaluated by the indirect method of Dual Energy Radiological Absortometry (DEXA) through the Prodigy® Lunar Bone Densitometry apparatus.

CONTACTS AND LOCATIONS:
Overall Officials: TATIANE AL SILVA, Ms, Principal Investigator — UFRN - Avenida Salgado Filho. S/N. Campus Central. Lagoa Nova. Rio Grande do Norte, Brazil
Locations (1):
- Universidade Federal Do Rio Grande Do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pannacciulli N, Salbe AD, Ortega E, Venti CA, Bogardus C, Krakoff J. The 24-h carbohydrate oxidation rate in a human respiratory chamber predicts ad libitum food intake. Am J Clin Nutr. 2007 Sep;86(3):625-32. doi: 10.1093/ajcn/86.3.625. PMID 17823426
- [Background] Kosmiski LA, Bessesen DH, Stotz SA, Koeppe JR, Horton TJ. Short-term energy restriction reduces resting energy expenditure in patients with HIV lipodystrophy and hypermetabolism. Metabolism. 2007 Feb;56(2):289-95. doi: 10.1016/j.metabol.2006.10.012. PMID 17224345
- [Background] Vassimon HS, de Paula FJ, Machado AA, Monteiro JP, Jordao AA Jr. Hypermetabolism and altered substrate oxidation in HIV-infected patients with lipodystrophy. Nutrition. 2012 Sep;28(9):912-6. doi: 10.1016/j.nut.2011.12.010. Epub 2012 Apr 13. PMID 22503533